CLINICAL TRIAL: NCT05490459
Title: Jewel Electrophysiology (EP) Lab Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Element Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-2038
Record Dates: First submitted 2022-07-27; First posted 2022-08-05 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-09

CONDITIONS: Sudden Cardiac Arrest
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Safety and Effectiveness
  Interventions: Device: Jewel Patch Wearable Cardioverter Defibrillator (P-WCD)

INTERVENTIONS:
Device: Jewel Patch Wearable Cardioverter Defibrillator (P-WCD) — Automatic external cardioverter defibrillator that monitors patients at risk for SCA and provides a therapeutic shock if needed.

SUMMARY:
Single arm open label evaluation of the Jewel Patch Wearable Cardioverter Defibrillator (P-WCD) defibrillation waveform in adult cardiac patients.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate safety and clinical effectiveness of the Jewel, using a single transthoracic defibrillation shock to terminate life-threatening VT or VF.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of both genders of at least 18 years of age.
2. Subjects who are scheduled for a standard EP clinical procedure where fast VT or VF may spontaneously occur or may be induced.

Exclusion Criteria:

1. Subjects who may require sterile access to the right upper pectoral or lower left torso regions during the planned EP procedure.
2. Subjects who have taken amiodarone in the past 3 months.
3. Subjects with an existing unipolar pacemaker.
4. Subjects who exhibit a left ventricular ejection fraction (LVEF) less than 20% (as assessed by techniques such as echocardiography, magnetic resonance imaging, or radionuclide angiography) within the last 6 months.
5. Subjects who have been diagnosed with heart failure (Class IV) or experienced an acute heart failure exacerbation within the previous 30 days.
6. Subjects who exhibit unstable angina.
7. Subjects with atrial fibrillation with contraindication to anticoagulation or improper anticoagulation management.
8. Subjects who are participating in an investigational study of a drug, biologic, or device not currently approved for marketing.
9. Subjects who are allergic to or have had a known adverse reaction to medical adhesives.
10. Subjects who have active skin breakdown, erythema, or other signs of infection in the pectoral or torso regions where the study device is applied.
11. Subjects with a lower abdomen circumference of less than 68.5 cm or greater than 142 cm.
12. Females who are pregnant or breastfeeding, or planning to be pregnant in the next 12 months.
13. Subjects who cannot provide or have diminished capacity to provide informed consent.
14. Any condition that an Investigator believes would interfere with the intent of the study or is not in the best interest of the patient.
15. Any patient that according to the Declaration of Helsinki is unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2024-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Petr Neužil, MD, PhD, FESC, Principal Investigator — Nemocnice na Homolce Hospital
Locations (1):
- Nemocnice Na Homolce Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chovanec M, Petru J, Hala P, Kralovec S, Thakkar AB, Mathews K, Dinger M, Ullery S, Eapen ZJ, Kumar UN, Neuzil P. First human safety and effectiveness study of defibrillation with a novel patch wearable cardioverter-defibrillator. Europace. 2024 Jul 2;26(7):euae189. doi: 10.1093/europace/euae189. PMID 39001864
- See also: Europace — https://pubmed.ncbi.nlm.nih.gov/39001864/

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Automatic external cardioverter defibrillator that monitors patients at risk for SCA and provides a therapeutic shock if needed.
Period: Overall Study
Arm/Group | Treatment
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 63.8 [28 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (kg/cm^2) [Mean (Full Range); unit: kg/cm^2] | 28.3 [20.2 to 36.9]

OUTCOME MEASURES:

1. Primary Outcome: Clinical Effectiveness of the Jewel
Description: The count of participants with successful single shock terminations of life-threatening VT or VF. (The endpoint would be achieved if the lower confidence limit exceeds the performance goal of 62% using a one-sided exact lower 97.4% confidence bound at one of three testing points.)
Time Frame: Immediately following defibrillation with the study device.
Population: Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 18
Participants | 16

ADVERSE EVENTS:
Time Frame: Enrollment to study exit following completion of EP clinical procedure (up to 24 hours).
Description: Adverse Events (AEs) defined as any untoward medical occurrence in a subject during the study.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the clinical trial or their parts shall not be published by Provider, Investigator, or other persons participating in the clinical trial shall not be disclosed to the general public without prior written consent of Sponsor. The Sponsor shall not refuses to grant consent without a reasonable cause.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT05490459/Prot_SAP_000.pdf